CLINICAL TRIAL: NCT05162326
Title: A Phase 1/2 Study of the Safety and Efficacy of BC-101 in Treatment of Nasolabial Fold Wrinkles Via Subcutaneous/Intradermal Injection
Brief Title: BC-101 in Treatment of Nasolabial Fold Wrinkles
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Cell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BC101-C01
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Nasolabial Fold Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BC-101 (Experimental): BC-101 will be injected at the dose of 0.1 mL per linear centimeter along the nasolabial fold, up to 2 mL in total volume for each side of the nasolabial folds.
  Interventions: Biological: BC-101

INTERVENTIONS:
Biological: BC-101 — Human umbilical cord tissue derived mesenchymal stem cells (hUC-MSC) suspension at concentration of 2, 4, or 6 million cells/mL.

SUMMARY:
This is an open-label, single-arm, dose-escalating study to evaluate the safety and tolerability of BC-101 administered via subcutaneous/intradermal injection in the treatment of moderate to severe nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are in general good health condition.
2. Subjects who have moderate to extremely deep bilateral nasolabial fold wrinkles, as documented by a score of 3 or greater on the six-point Evaluator Wrinkle Severity Assessment scale (0-5).
3. Subjects who are dissatisfied with both nasolabial fold wrinkles based on a score of -1 or -2 on the Subject Wrinkle Assessment Scale (-2 to +2).
4. Subjects who voluntarily adhere to the research procedures and ensure good compliance during the research period.
5. Subjects who fully understand the research nature of this study and sign the informed consent.

Exclusion Criteria:

1. Subjects who have an active cutaneous infection on the face.
2. Subjects with existing malignant neoplasm.
3. Subjects with persistent pre-cancerous lesions (e.g., actinic keratosis).
4. Subjects who have active dermal diseases, inflammation, or any related disease.
5. Subjects who have cosmetic or surgical treatment on nasolabial fold area in 3 months before the study (including laser, chemical peels, fillers, botulinum toxin).
6. Subjects who are pregnant, breastfeeding, or whose urinary pregnancy test is positive before participation in the study.
7. Subjects who are allergic to low-molecular-weight heparin sodium or human albumin.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of any treatment-emergent adverse events | 12 weeks after injection

SECONDARY OUTCOMES:
Changes in wrinkle severity assessment from baseline | 6 weeks, 12 weeks and 26 weeks after injection
  Each of the bilateral nasolabial fold wrinkles at rest will be evaluated using the 6-point ordinal Lemperle Wrinkle Severity Scale.